CLINICAL TRIAL: NCT03704194
Title: Adapted Lifestyle-integrated Functional Exercise Program for Older Adults in Under Resourced Communities: A Pilot Study
Brief Title: Adapted Lifestyle-integrated Functional Exercise Program for Medically Underserved Older Adults
Acronym: LiFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201807067
Record Dates: First submitted 2018-09-18; First posted 2018-10-12 (Actual); Results first posted 2020-07-28 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Accidental Fall
Keywords: falls; exercise program; medically underserved

STUDY DESIGN:
Intervention Model Description: randomized controlled feasibility trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted LiFE (Experimental): Participants in the Adapted LiFE group learns to imbed 19 exercise activities (7 balance and 12 lower extremity muscle strength activities) into daily routines. An Occupational Therapy practitioner conducts 7 in-home visits over 12 weeks and a follow phone call a month after the last in-home visit.
  Interventions: Behavioral: Adapted LiFE
- Attention control (Sham Comparator): Participants in the attention control group will learn gentle stretch exercise. An Occupational Therapy practitioner conducts 7 in-home visits over 12 weeks and a follow phone call a month after the last in-home visit.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: Adapted LiFE — The standardized components include presenting the Adapted LiFE user manual to participants, and teach participants to embed the exercise activities in their daily routine with the LiFE activity calendar.
  Arms: Adapted LiFE
Behavioral: Attention control — Attention will be provided to the control group to ensure they experience the same effects of time and attention but no effect on the outcome of interest.
  Arms: Attention control

SUMMARY:
This study will test the feasibility of a study design for the Adapted Lifestyle-integrated Functional Exercise (LiFE) program for medically underserved older adults and to explore factors related to implementation. A feasibility trial will be conducted with a total of 16 participants. The control group will receive flexibility exercise program as attention control.

DETAILED DESCRIPTION:
This study will test the feasibility the Adapted Lifestyle-integrated Functional Exercise (LiFE) program among medically underserved older adults. Sixteen medically underserved older adults will be recruited in the study and randomized to Adapted LiFE or attention control group (flexibility exercise program). Process outcomes and preliminary outcomes will be collected to determine feasibility and preliminary efficacy. Process outcomes such as reach, acceptance, adherence, fidelity, and safety will also be collected throughout the study. Preliminary efficacy outcomes include habit formation, balance, muscle strength will be collected at baseline and at immediately after intervention is completed.

ELIGIBILITY:
Inclusion Criteria:

* (1) age 70 or older;
* (2) live independently;
* (3) live in a medically underserved/health professional shortage area;
* (4) self-report two falls or one injurious fall.

Exclusion Criteria:

* (1) Short Blessed Test score ≥8, indicating cognitive impairment consistent with dementia;
* (2) inability to stand independently with a walking device;
* (3) having a serious health condition with a physician's order where exercise is contraindicated.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stark, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
The results are not published yet.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adapted LiFE | Attention Control
Started | 8 | 9
Completed | 8 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapted LiFE | Attention Control | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.0 (4.9) | 77.9 (6.7) | 77.0 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  sex: Female | 6 | 6 | 12
  sex: Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Berg Balance Scale (BBS)
Description: The Berg Balance Scale (BBS) is a 14-item assessment of static and dynamic balance. Performance quality, time, and assistance required are rated on a scale of 0-4 based on pre-specified criteria. Total scores range from 0-56, with a score of 45 or below indicating high risk of falls.
Time Frame: Baseline and 12 weeks
Population: Participants who completed the intervention were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adapted LiFE | Attention Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Pre-test | 40.63 (10.17) | 35.25 (11.52)
  Post-test | 38.38 (12.59) | 35.88 (9.85)

2. Secondary Outcome: The Self-Reported Habit Index (SRHI)
Description: The Self-Reported Habit Index (SRHI) is a 12-item assessment assesses habit exercise strength, frequency, relevance to self-identity, and automaticity. Items are self-rated with a seven-point Likert scale (1=strongly disagree, 7= strongly agree). Total score range from 12 to 84, where higher scores indicate stronger the habit is.
Time Frame: Baseline and 12 weeks
Population: Participants in the treatment group were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adapted LiFE
Number analyzed (Participants) | 8
score on a scale
  Pre-test | 47.50 (21.67)
  Post-test | 57.13 (19.26)

3. Secondary Outcome: The Activities-specific Balance Confidence Scale (ABC)
Description: The Activities-specific Balance Confidence Scale (ABC) is 16-item self-report measure in which participates rate their balance confidence for performing activities. Each item is rated on a 0-100 scale (0= no confidence, 100 = complete confidence). A final score is the average of all items ( range from 0 to 100).
Time Frame: 12 weeks
Population: All participants who completed the interventions were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adapted LiFE | Attention Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Pre-test | 60.77 (20.83) | 52.46 (22.26)
  Post-test | 60.63 (21.57) | 60.7 (12.94)

4. Secondary Outcome: The Short Physical Performance Battery (SPPB)
Description: The Short Physical Performance Battery-Balance Test (SPPB) assess balance and mobility with three subtests (score range: 0 to 4): standing balance, three-meter gait speed, and five repetitions of sit-to-stand motion. Total score are sums of subtest scores ranging from 0 (worst performance) to 12 (best performance).
Time Frame: Baseline and 12 weeks
Population: Participants who completed the interventions were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adapted LiFE | Attention Control
Number analyzed (Participants) | 8 | 8
score on a scale
  Pre-test | 6.38 (2.83) | 5.25 (2.87)
  Post-test | 5.25 (3.01) | 5.38 (2.20)

5. Secondary Outcome: Center of Pressure (CoP) Path (cm)
Description: Center of Pressure (Cop) is measured by a balance board system BtracKS. Participant stands on the balance board in 4 posture in three 30-second trials for each posture: hip-width stand (HS), hip-width stand with eyes closed (HSEC), narrow stand (NS), narrow stand with eyes closed (NSEC). Trajectory and mean velocity of CoP in each postures are calculated to represent static balance. Larger trajectory or velocity indicates lower static balance.
Time Frame: Baseline and 12 weeks
Population: Participants who completed the interventions were included in the analysis.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Adapted LiFE | Attention Control
Number analyzed (Participants) | 8 | 8
cm
  HS CoP Mean distance (cm) Pre-test | 0.59 (0.13) | 0.67 (0.32)
  HS CoP Mean distance (cm) Post-test | 0.68 (0.16) | 0.61 (0.19)
  HSEC CoP Mean distance (cm) Pre-test | 0.59 (0.13) | 0.69 (0.29)
  HSEC CoP Mean distance (cm) Post-test | 0.68 (0.16) | 0.72 (0.30)
  NS CoP Mean distance (cm) Pre-test | 0.82 (0.09) | 0.71 (0.17)
  NS CoP Mean distance (cm) Post-test | 1.03 (0.43) | 0.83 (0.32)
  NSEC CoP Mean distance (cm) Pre-test | 1.13 (0.24) | 0.99 (0.40)
  NSEC CoP Mean distance (cm) Post-test | 1.39 (0.51) | 1.12 (0.54)

6. Secondary Outcome: Center of Pressure (CoP) Velocity (cm/s)
Description: Center of Pressure (Cop) mean velocity (cm/s) is measured by a balance board system BtracKS. Participant stands on the balance board in 4 posture in three 30-second trials for each posture: hip-width stand (HS), hip-width stand with eyes closed (HSEC), narrow stand (NS), narrow stand with eyes closed (NSEC). Larger velocity indicates a lower static balance.
Time Frame: Baseline and 12 weeks
Population: Participants who completed the interventions were included in the analysis.
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Adapted LiFE | Attention Control
Number analyzed (Participants) | 8 | 8
cm/s
  HS CoP Mean velocity (cm/s) Pre-test | 2.38 (1.05) | 1.96 (0.55)
  HS CoP Mean velocity (cm/s) Post-tes | 2.59 (1.52) | 1.96 (0.74)
  HSEC CoP Mean velocity (cm/s) Pre-test | 3.22 (2.03) | 2.89 (1.11)
  HSEC CoP Mean velocity (cm/s) Post-test | 4.01 (3.48) | 3.02 (1.12)
  NS CoP Mean velocity (cm/s) Pre-test | 3.18 (1.31) | 2.93 (0.75)
  NS CoP Mean velocity (cm/s) Post-test | 3.88 (2.20) | 2.45 (1.05)
  NSEC CoP Mean velocity (cm/s) Pre-test | 4.55 (1.88) | 4.21 (2.30)
  NSEC CoP Mean velocity (cm/s) Post-test | 5.05 (2.38) | 4.30 (2.53)

7. Secondary Outcome: Lower Extremity Muscle Strength
Description: Lower extremity muscle strength of hip and knee are measured by a dynamometer.
Time Frame: Baseline and 12 weeks
Population: Participants who completed the interventions were included.
Measure: Mean (Standard Deviation); unit: pound
Arm/Group | Adapted LiFE | Attention Control
Number analyzed (Participants) | 8 | 8
pound
  Hip flexors (right limb) Pre-test | 18.11 (4.37) | 19.86 (8.95)
  Hip flexors (right limb) Post-test | 18.73 (12.55) | 21.58 (15.75)
  Hip flexors (left limb) Pre-test | 17.10 (4.94) | 15.97 (7.67)
  Hip flexors (left limb) Post-test | 19.79 (13.23) | 19.25 (8.70)
  Knee flexors (right limb) Pre-test | 23.83 (2.96) | 24.15 (8.91)
  Knee flexors (right limb) Post-test | 16.48 (9.51) | 18.65 (8.22)
  Knee flexors (left limb) Pre-test | 21.34 (4.47) | 23.40 (6.66)
  Knee flexors (left limb) Post-test | 15.01 (8.61) | 19.1 (8.77)
  Knee extensors (right limb) Pre-test | 25.38 (6.90) | 27.38 (7.53)
  Knee extensors (right limb) Post-test | 22.62 (9.18) | 27.15 (10.84)
  Knee extensors (left limb) Pre-test | 23.25 (8.06) | 26.56 (6.84)
  Knee extensors (left limb) Post-test | 21 (9.19) | 26.81 (11.15)

8. Other Pre Specified Outcome: Recruitment and Retention Rate Are Documented by Therapist Logs
Description: The status of each potential participant we contacted is documented in an electronic therapist log. Treatment and control groups share the same recruitment rate since randomization took place after enrollment, and the two groups were not recruited separately. Recruitment rate will be measured by the percentage of participants successfully enrolled in the study. Retention rate is calculated by the number of participants completed divided by the number of participants enrolled. Retention rate is calculated by the number of participants completed divided by the number of participants enrolled.
Time Frame: 16 weeks
Population: Among 39 potentially eligible participants, 16 successfully enrolled. The 16 enrolled participants were randomized to treatment (n=8) and control (n=8)groups, and all completed the intervention and one-month follow-up, which resulted in a 100% retention rate.
Measure: Number; unit: percentage of participants
Arm/Group | Attention Control | Adapted LiFE
Number analyzed (Participants) | 8 | 8
percentage of participants
  Recruitment rate | 42.02 | 42.02
  Retention rate | 100 | 100

9. Other Pre Specified Outcome: Acceptance of the Intervention Programs is Measured by a Question.
Description: A question, "Are you satisfied with the program?," using a seven-point Likert scale from one (very unsatisfied) to seven (very satisfied) is used to represent acceptance. Score range: 1-7. Higher values indicate higher satisfaction.
Time Frame: 12 weeks
Population: Participants completed treatment intervention were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adapted LiFE
Number analyzed (Participants) | 8
score on a scale | 6.88 (0.35)

10. Other Pre Specified Outcome: Adherence Rate is Documented by LiFE Activity Calendar
Description: Participants in the treatment group documents their exercise activities in the LiFE activity calendar. Adherence rate is defined as the average percentage of exercise activities achieved during the intervention period.
Time Frame: 12 weeks
Population: Participant in the treatment group.
Measure: Mean (Standard Deviation); unit: percentage of achieved exercise activity
Arm/Group | Adapted LiFE
Number analyzed (Participants) | 8
percentage of achieved exercise activity
  Session 1 | 79 (33)
  Session 2 | 87 (12)
  Session 3 | 73 (23)
  Session 4 | 76 (35)
  Session 5 | 73 (35)
  Session 6 | 74 (34)
  Session 7 | 51 (46)

11. Other Pre Specified Outcome: Fidelity is Documented by a Visit-by-visit Checklist
Description: Therapists in both treatment and control group complete a checklist after every visit. The checklist consist of pre-determined key activities. The number of delivered key activities divided by the number of planned key activities in all visits calculates a fidelity score.
Time Frame: 12 weeks
Population: Participants completed the interventions were included.
Measure: Mean (Standard Deviation); unit: percentage of treatment delivery
Arm/Group | Adapted LiFE | Attention Control
Number analyzed (Participants) | 8 | 8
percentage of treatment delivery | 100 (0) | 100 (0)

12. Other Pre Specified Outcome: Adverse Events
Description: Safety of the program will be evaluated by the number of adverse events documented throughout the study duration.
Time Frame: 16 weeks
Population: Participants completed the interventions were included.
Measure: Mean (Standard Deviation); unit: counts of adverse events
Arm/Group | Adapted LiFE | Attention Control
Number analyzed (Participants) | 8 | 8
counts of adverse events | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through a 16-week period when a participant was enrolled in the study.
Arm/Group | Adapted LiFE | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT03704194/Prot_SAP_000.pdf